CLINICAL TRIAL: NCT00576485
Title: Spherical Aberration and Contrast Sensitivity in Eyes Implanted With Aspheric and Spherical Intraocular Lenses: Clinical Comparative Study
Brief Title: Spherical Aberration and Contrast Sensitivity in IOLs
Acronym: IOLs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Patrick Frensel de Moraes Tzelikis, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 490/06; ETIC490/06
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2007-12

CONDITIONS: Cataract; Signs and Symptoms; Pseudophakia; Lens Diseases
Keywords: Cataract; Intraocular lens; Spherical aberration; Contrast sensitivity
MeSH Terms: conditions — Cataract; Signs and Symptoms; Pseudophakia; Lens Diseases | interventions — Cataract Extraction; Lens Implantation, Intraocular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cataract surgery and implantation of a spherical intraocular lens
  Interventions: Procedure: Cataract surgery and intraocular lens implantation
- 2 (Experimental): Cataract surgery and implantation of a spherical intraocular lens
  Interventions: Procedure: Cataract surgery and intraocular lens implantation

INTERVENTIONS:
Procedure: Cataract surgery and intraocular lens implantation — Cataract surgery and implantation of an intraocular lens

SUMMARY:
Purpose: To determine whether implantation of an intraocular lens (IOL) with a modified anterior aspheric surface results in reduced spherical aberration and improved contrast sensitivity after cataract surgery.

Design: Prospective, comparative, interventional case series.

Methods: In an intraindividual randomized prospective study of 25 patients with bilateral cataract, an IOL with a modified anterior surface (Tecnis Z9001, AMO- Group 1) was compared with biconvex lens with spherical surfaces (ClariFlex®, AMO- Group 2). Ocular aberrations for a 5.0 mm pupil and 6.0 mm pupil were measured with Hartmann-Shack aberrometer. Quality of vision was measured by visual acuity and contrast sensitivity under mesopic and photopic conditions. All patients were followed for 3 months.

DETAILED DESCRIPTION:
With improvement in the quality of life and the resulting expansion of the elderly population, the prevalence of cataract cases will continue to rise. The population is on average older, and the environment has become more demanding for older people, who therefore need to regain excellent quality of vision. Advances in both IOL and phacoemulsification technology have enable cataract surgery to evolve from a procedure concerned with the safe removal of the cataract to a procedure refined to achieve the best possible postoperative refractive result.

Snellen visual acuity insufficiently describes the quality of the eye's optics before and after cataract surgery. 1-3 Multiple scientific studies have demonstrated that contrast sensitivity represents a robust indicator of functional vision. 4-7 The contrast sensitivity function, measured under varying conditions of luminance and glare, establishes the limits of visual perception across the spectrum of spatial frequencies.

Studies have demonstrated a nearly linear decline in image quality with age, suggesting a significant increase in the optical aberrations in the eye over time. 8-9 Advances in wavefront technology have opened a new door to the measurement of ocular aberrations. 9-10 Also, this technology allowed the development of a new type of IOL designed to compensate for the positive spherical aberration of the cornea, which is one of the most important aberrations contributing to visual deterioration of the pseudophakic eye. 11-14 Based on these findings, the approach to compensate for increasing spherical aberration in older eyes is to develop an IOL that introduces negative spherical aberration into the system. Such an IOL, the Tecnis Z9001® IOL (Model Z9001, Advanced Medical Optics, Santa Ana, CA), has been developed by AMO. This is a polysiloxane foldable 3-piece IOL, with anterior aspheric surface (negative spherical aberration) designed to decrease the total amount of ocular spherical aberration after cataract surgery.7

The purpose was to determine whether implantation of an intraocular lens (IOL) with a modified anterior aspheric surface results in reduced spherical aberration and improved contrast sensitivity after cataract surgery.

Patients and Methods

This double-blind prospective randomized study included patients with age-related cataract, no indication of existing ocular pathology, unsatisfactory correction with glasses and less than 2.50 diopters (D) of topography cylinder. Patients were offered the opportunity to be part of a clinical trial in which they would be allocated to have cataract surgery with implantation of aspherical or spherical IOL. Patients were randomized to receive a Tecnis Z9001 aspheric IOL in one eye and a ClariFlex spheric IOL in the fellow eye. To protect patient safety, after the first eye surgery, they were asked whether they wished to have the same lens type implanted in the second eye. Written informed consent was obtained from all patients before surgery and the study was approved by the local ethics committee. Exclusion criteria were previous ocular surgery, central endothelial cell count less than 1800 cells/mm2, glaucoma or intraocular pressure greater than 21 mmHg, amblyopic eyes, retinal abnormalities, diabetes mellitus, steroid or immunosuppressive treatment, and connective tissue diseases.

The selected lenses used in this study were the Tecnis Z9001® (Model Z9001, Advanced Medical Optics, Santa Ana, CA) and the ClariFlexTM (Advanced medical Optics, Santa Ana, CA) (Table 1). Eyes in Group 1 (n=25) received the Tecnis Z9001® (Model Z9001) and eyes in Group 2 (n=25) received the ClariFlexTM (Table 1).

The Holladay formula was used to calculate the IOL power when there was a short axial length (< 22.0 mm) and the SRK/T formula was used when there was an average axial length (≥ 22.0 mm). The A-constant used was 119.1 for the Tecnis Z9001 IOL and 118.0 for the ClariFlex IOL. Axial length was measured with the IOL Master (Carl Zeiss Meditec AG), and the targeted postoperative refractive error was 0.0.

Preoperative and postoperative evaluation included uncorrected distance visual acuity (UCDVA), best corrected visual acuity (BCVA), spherical equivalent (SE), slitlamp biomicroscopy, applanation tonometry, fundus examination, B-scan biometry, specular microscope and corneal topography. Topography was performed in all patients using the EyeSys unit (Version 3.03; EyeSys Technologies, Houston, Texas). The corneal endothelial cell count was also recorded for all eyes (noncontact specular microscope, NonCon Robo, Konan). The visual acuity measurements were recorded with logMAR UCDVA and BCVA. Clinical data were collected preoperatively and 1 and 3 months postoperatively for each eye.

All patients were operated in the same fashion by the same surgeon. All patients received topical anesthesia by lidocaine 2% gel before surgery. A 2.75 mm self-sealing clear cornea incision was made on the temporal side. Viscoelastic solution of sodium hyaluronate 3% and chondroitin sulfate 4% (Viscoat®) was used to reform and stabilize the surgical planes and protect the endothelium. A 5.00 to 5.25 mm continuous curvilinear capsulorhexis was initially performed with a 26-gauge needle and completed with forceps. The nucleous was removed without intraoperative complications such as posterior capsule rupture. Phacoemulsification was performed using the Infinite (Alcon Surgical) or Sovereign machine (Allergan Surgical). All IOLs were inserted in the capsular bag with the injector system. The viscoelastic material was completely removed at the end of the procedure. No sutures were used in any case. After 1 week the patient had the fellow eye operated. Postoperative medication included moxifloxacin (Vigamox®) or gatifloxacin (Zymar®) 4 times a day for 2 weeks, 0.1% diclofenaco sodium (Voltaren) 3 times a day for 4 weeks and steroid (Predfort) eyedrops 4 times a day for 6 weeks. Postoperative follow-up was 1 day, 1 and 3 months.

Postoperative evaluations were performed at 1 day, 1 month, and 3 months. At 1 month and 3 months, visual acuity, refraction, contrast sensitivity (CSV-1000 HGT, Vector Vision Inc.), and wavefront analysis with the Zywave aberrometer (Bauch & Lomb, Rochester, New York) were performed.

Contrast sensitivity was measured using the CSV-1000 HGT testing instrument (Vector Vision Inc.), which presents a translucent chart divided into 4 cycles with spatial frequencies of 3, 6, 12, and 18 cycles per degree (cpd). The background illumination of the translucent chart does not depend on room lighting; rather, it is provided by a fluorescent luminance source of the instrument and is automatically calibrated to 85 candelas/m2. All measurements were obtained under mesopic (5 cd/m2) and photopic (85 cd/m2) conditions. Each cycle contains 17 round patches that are 1.5 inches in diameter. The first patch has a high-contrast grating and presents the sample. The test patches are arranged in 2 rows with 8 levels of contrast. The levels decreased from left to right along the row in a logarithmic fashion in 0.17 log units for steps 1 through 3 and 0.15 log units for steps 3 through 8. The examinations were performed unilaterally at a distance of 2.5 m with best corrected visual acuity (BCVA) and an undilated pupil. All measurements were conducted under the same conditions by an examiner who was unaware of the type of IOL implanted.

Wavefront analysis was performed by the Zywave aberrometer. The Zywave aberrometer uses the Hartmann-Shack method of analysis of the outgoing wavefront that measures up to fifth-order Zernike aberrations, including coma, trefoil, and spherical aberrations.

For statistical analysis of visual acuity, logarithm of minimum angle of resolution (logMAR) acuity values were used. Similarly, the recorded contrast sensitivity values were transformed into log values as described by Vector Vision. All data analyses were performed using SPSSX statistical programs (SPSS Inc, Chicago, IL). The 2 IOLs were compared between eyes intraindividually. The analysis was based on a non-normal distribution of the data. The nonparametric Mann-Whitney U test was used to compare data between the 2 IOL groups. A P value less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract
* No indication of existing ocular pathology
* Unsatisfactory correction with glasses and
* Less than 2.50 diopters (D) of topography cylinder.

Exclusion Criteria:

* Previous ocular surgery
* Central endothelial cell count less than 1800 cells/mm2
* Glaucoma or intraocular pressure greater than 21 mmHg
* Amblyopic eyes
* Retinal abnormalities
* Diabetes mellitus
* Steroid or immunosuppressive treatment, and
* Connective tissue diseases

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-02; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To determine whether implantation of an intraocular lens (IOL) with a modified anterior aspheric surface results in reduced spherical aberration and improved contrast sensitivity after cataract surgery | within the first 30 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Patrick F Tzelikis, MD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Federal University of Minas Gerais - Sao Geraldo Eye Hospital, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Derived] Tzelikis PF, Akaishi L, Trindade FC, Boteon JE. Spherical aberration and contrast sensitivity in eyes implanted with aspheric and spherical intraocular lenses: a comparative study. Am J Ophthalmol. 2008 May;145(5):827-33. doi: 10.1016/j.ajo.2007.12.023. Epub 2008 Mar 4. PMID 18291345